CLINICAL TRIAL: NCT01703650
Title: Evaluation of Diagnostic Efficacy of Perfusion CT Using Wide Detector for Staging and Response Prediction After Chemotherapy in Pancreatic Cancer
Brief Title: Role of Perfusion CT in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: SNUH_ISS_2012
Record Dates: First submitted 2012-10-06; First posted 2012-10-10 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Adenocarcinoma, Pancreas; Neuroendocrine Carcinoma of Pancreas
Keywords: CT; pancreas adenocarcinoma; RECIST; perfusion
MeSH Terms: conditions — Adenocarcinoma | interventions — iopromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Resectable pancreas cancer: patients with resectable pancreas adenocarcinoma or neuroendocrine tumor underwent perfusion CT after intravenous iopromide administration
  Interventions: Drug: iopromide; Procedure: CT
- Locally advanced Pancreas cancer: Patients with locally advanced pancreas cancer underwent perfusion CT after intravenous iopromide administration before and after chemotherapy.
  Interventions: Drug: iopromide; Procedure: CT

INTERVENTIONS:
Drug: iopromide — 1. iopromide (370mgI/mL) enhanced perfusion CT will be performed within 14 days of operation.
  2. In patients who are planned to receive chemotherapy, iopromide enhanced perfusion CT was performed twice; within 14 days before starting 1st cycle and within 14 days after finishing 2nd cycle.
  3. iopromide (370mgI/mL) will be administered intravenously with an amount of 30mL (body weight[BW] <50kg) or 35 mL (50kg ≤BW <70kg) or 40 mL (70 kg≤BW <90kg) or 50 mL (90≤BW), followed by saline infusion (30mL).
  4. Injection rate is as follows; 6.0mL/sec if BW is <50kg, 7.0 mL/sec if BW is 50kg≤and <70kg, 8.0 mL/sec if BW is 70≤and<90kg and 9.0mL/sec if BW is 90kg≤.
  Other Names: Ultravist® (370mgI/mL)
Procedure: CT — 1. Perfusion CT will be performed by using a 320 channel MDCT
  2. Patients are requested for fasting for at least 8 hours before CT scan.
  3. Patients are requested for doing shallow breathing as slow as possible and wide strap is applied during CT scan.
  4. Scan range is limited to the whole pancreas and it focuses to the pancreas tumor lesion.
  5. During perfusion CT, 19 phases (ten phases with two seconds interval and six phases with three seconds interval and three phases with five seconds interval) are obtained in fifty three seconds.
  6. ADIR 3D and SURE EXPOSURE 3D are applied during perfusion CT to minimize radiation dose.

SUMMARY:
The purpose of this study is

1. to determine whether the perfusion parameters in the normal pancreas and the pancreas cancer (adenocarcinoma or neuroendocrine tumor) are different on perfusion CT
2. to determine whether initial perfusion parameters as well as perfusion parameter change in pancreas adenocarcinoma before and after chemotherapy are different between chemotherapy response group (CR, PR according to RECIST 1.1) and non response group (SD, PD according to RECIST 1.1).

DETAILED DESCRIPTION:
1. Performance of preoperative perfusion CT for preoperative staging is assessed by comparing with operative finding and histologic disease staging
2. Estimation of initial or change of pancreas cancer perfusion parameters and whether those can provide cut-off value for predicting response of chemotherapy in patients with pancreas adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* patients who are older than eighteen years
* patients in whom operation and preoperative computed tomography are scheduled for resectable pancreas adenocarcinoma or pancreas neuroendocrine tumor
* patients in whom chemotherapy is scheduled for histologically confirmed pancreas adenocarcinoma
* patients in whom chemotherapy is planned for highly suspicious pancreas adenocarcinoma on imaging workup
* patients who agree with the study and whose informed consent is obtained.

Exclusion Criteria:

* patients who are younger than eighteen years old
* patients in whom previously radiation therapy was performed and the RTx field includes pancreas
* patients with recurred pancreas adenocarcinoma
* patient who are pregnant or nursing patients
* patients with renal failure (GFR<30mL/min)
* patients with history of malignancy, except malignancy is in complete remission after operation or iodine therapy for at least five years)
* patients with hypersensitivity for iodine or contrast media or other causes of contraindication of contrast-media enhanced CT scan
* Any other condition which, in the opinion of the Investigator, would make the patient unsuitable for enrollment or could interfere with the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resectable pancreas tumor group patients with resectable pancreas adenocarcinoma or neuroendocrine tumor
  Locally advanced pancreas tumor group Patients with locally advanced pancreas cancer
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the correlation between the initial perfusion parameters of the tumor and response of the chemotherapy | after 6 cycles of the planned chemotherapy
  Initial perfusion parameters (blood volume, blood flow and permeability) are compared between CTx-responder and non-responders after 6 cycle of the scheduled chemotherapy, using RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Correlation between change of perfusion parameters and the chemotherapy response | after 6 cycles of the chemotherapy
  Perfusion parameters (blood volume, blood flow, and permeability) change between initial perfusion CT and second perfusion CT (which is taken after 2 cycle of the CTx) are compared between CTx-responder and non-responder after finishing 6 cycles of CTx according to RECIST 1.1 criteria.
Perfusion parameters among different pancreas tumors | within 2 months after finishing enrollment
  Perfusion parameters (blood volume, blood flow and permeability) are compared among the different types of the pancreas tumors to investigate perfusion parameters can help characterization of the tumors.
comparison of perfusion parameters among the pancreas tumors and parenchyma | within three weeks before pancreas tumor surgery
  blood volume, blood flow and permeability are compared between the tumor and the pancreas parenchyma.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No